CLINICAL TRIAL: NCT01329601
Title: Effect of the Stage Specific Cognitive Intervention Program on Functional Cortical Activation in Alzheimer's Disease
Brief Title: Effect of Cognitive Intervention in Alzheimer's Disease (AD) on Functional Cortical Networks in fMRI
Acronym: ECIF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Collaborators: DZNE, German Center for Neurodegenerative Disorders, Germany (Unknown)
Responsible Party: Stefan Teipel, Department of Psychiatry, University Rostock
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Int_HRO_1
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-01

CONDITIONS: Dementia of the Alzheimer Type
Keywords: cognitive training; Alzheimer disease; tertiary prevention
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Intervention (Experimental): StaCog intervention to improve cognitive performance and activities of daily living in AD and MCI
  Interventions: Behavioral: StaCog, stage specific cognitive Intervention
- Booklet-based training (Active Comparator): Home based training of episodic memory using paper-pencil exercizes
  Interventions: Behavioral: booklet based training

INTERVENTIONS:
Behavioral: StaCog, stage specific cognitive Intervention — StaCog intervention to improve cognitive performance and activities of daily living in AD and MCI
  Other Names: Cognitive rehabilitation
  Arms: Cognitive Intervention
Behavioral: booklet based training — Home based training of episodic memory using paper-pencil exercizes
  Other Names: Active behavioural control
  Arms: Booklet-based training

SUMMARY:
The study aims to detect the effect of a structured cognitive rehabilitation program, teh stage specific intervention STACog, on cognitive performance and functional activation in fMRI in a group of patients with mild cognitive impairment and dementia due to Alzheimer's disease compared to a waiting group control sample. Baseline performance in cognitive tests and fMRI will further be assessed compared to healthy control subjects.

DETAILED DESCRIPTION:
Subject of the proposed project is to offer based on existing theoretical principles and methods stage-related, reproducible, relevant to everyday life group training in German for people with aMCI and slightly severe AD and compared with a - in terms of goal variables - to be less effective prestigious intervention . It is believed that the "active treatment" - in the intervention group, the overall level of functioning can longer be maintained and that positive transfer effects on non-cognitive level - to achieve and cognitive level - here at nationals. In addition, information is expected that the conversion rate of people with dementia and aMCI cut to a further loss of independence in humans can be delayed slightly with severe AD. The project aims to provide data to estimate the effect sizes of intervention can be determined on the basis of group size and duration of ongoing investigations.

Involving functional imaging measures, the intervention study, an adequate platform for the detection of intervention effects on neurobiological basis using fMRI dar. Here, the cerebral blood flow in specific activation as a measure of neuronal and synaptic activity and integrity both in cross-section of a subsample of healthy elderly people studied determined and changes in cerebral activity patterns in people with severe AD, aMCI or slightly in comparison pre-/post interventions. There are detectable much earlier in the pathogenesis of functional changes as structural, using fMRI, the study is to make a significant contribution to prove whether a modular cognitive intervention altered neural and synaptic activity and whether this change is accompanied by an improvement in cognitive performance.

A complete and proven effectiveness of cognitive group training could make a significant contribution that people with MCI and severe AD easily submit their own initiative mental condition, and add itself to sustain the intellectual, emotional and social potential. As a long-term perspective, the results for the optimization of cognitive intervention programs and continue to implement the organizations of the open and contribute stationary the elderly and specialized medical facilities and other medical facilities.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Mild Cognitive Impairment, Amnestic type (single domain) according to Petersen criteria or a low grade AD according to ICD-10/NINCDS-ADRDA

Exclusion Criteria:

* Major depression
* severe visual and acoustic impairment
* severe physical impairments
* known malignancy
* laboratory elevated inflammatory markers (ESR, CRP, leukocytes)
* stroke
* brain trauma
* epilepsy
* previous participation in a memory training
* patients receiving drug treatment (antidepressants, neuroleptics, anti-dementia, other brain performance enhancing drugs) at least three months prior to study initiation for the duration of the project are at a stable dosage

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
California Verbal Learning Test | Detecting changes between two different time points (baseline and 6 months)
  Cognitive test for episodic memory

SECONDARY OUTCOMES:
functional cortical activity in fMRI | Detecting changes between two different time points (baseline and 6 months)
  Measure of cortical activation during n-back letter recognition with emotional modulation

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J. Teipel, Prof. Dr., Principal Investigator — Klinik für Psychiatrie und Psychotherapie, Universitätsklinikum Rostock
Locations (1):
- Department of Psychiatry, University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany